CLINICAL TRIAL: NCT05898477
Title: Describing Treatment Outcomes and Responses in Lymphoma-associated Hemophagocytic Lymphohistiocytosis
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gaurav Goyal, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300010383
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma; Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Lymphoma; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophagocytic lymphohistiocytosis (HLH) Patients

SUMMARY:
The purpose of the study is to describe Hemophagocytic lymphohistiocytosis (HLH) in patients with lymphoma to identify possible therapeutic strategies to improve overall survival of the patients with lymphoma associated hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
Retrospective, multi-institutional study focused on describing the clinical features, laboratory parameters, treatments, and outcomes among individuals presenting with HLH in the setting of a lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma that are fulfilling at least one of the following:

A. Meeting 5 of 8 HLH-2004 diagnostic criteria OR B. Are OHI index positive (sCD25>3,900 U/mL and ferritin>1,000 ng/mL)

Exclusion Criteria:

* Patients developing HLH> 1 month after lymphoma diagnosis (for aggressive lymphomas)
* Patients with incomplete treatment and response documentation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of Hemophagocytic lymphohistiocytosis (HLH)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To determine the factors predicting 180 days overall survival of patients with cancer that are HLH-2004/OHI+ | The participant's survival would be assessed at 180 days from the malignancy diagnosis
  The investigators will gather data on different treatments received, time to treatment, and other factors and determine which is associated with survival.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Goyal, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States